CLINICAL TRIAL: NCT03417440
Title: A Smartphone Application to Improve Physical Activity in Underactive Older Adults
Brief Title: A Smartphone App to Improve Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institute on Aging (NIA) (NIH); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Stacey L. Schepens Niemiec, Assistant Professor of Research, University of Southern California
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Other
Other Study IDs: HS-16-00670; R21AG052838 (NIH)
Record Dates: First submitted 2018-01-24; First posted 2018-01-31 (Actual); Results first posted 2022-11-21 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-10

CONDITIONS: Sedentary Lifestyle
Keywords: smartphone app, physical activity, older adults
MeSH Terms: conditions — Sedentary Behavior; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Multiphase Optimization Strategy (MOST) is a recent methodology for optimizing multi-component interventions prior to performing more comprehensive testing in large RCTs. The Most Framework includes 5 steps: (1) Establish theoretical model; (2) Identify individual intervention components; (3) Conduct experiment to examine individual components; (4) Assemble beta intervention package; and (5) Confirm efficacy of optimized intervention. To our knowledge, only two prior studies have used MOST to refine a complex app with physical activity elements and disentangle the relative efficacy of specific features within a larger suite.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Study measures (apart from accelerometry, Health-ITUES, and usage data-see below) will be administered by a condition-blind tester at a study site at baseline and post-intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- PA App+ On Your Feet+ CoachMe+ Proof Pos (Other): Participants in this arm will use a basic physical activity (PA) tracker app in conjunction with the following 3 features: (1) "On Your Feet" (sedentary activity monitoring with motivational messaging and peer suggestions); (2) "Coach Me" (tailored messaging to increase the intensity level of everyday activities and overcome barriers); and (3) "Proof Positive" (explicit and implicit messaging to promote positive aging views).
  Interventions: Other: Physical Activity (PA) Tracker App; Other: On Your Feet; Other: Coach Me; Other: Proof Positive
- PA App + On Your Feet + Coach Me (Other): Participants in this arm will use a basic physical activity (PA) app in conjunction with the following 2 features: (1) "On Your Feet" (sedentary activity monitoring with motivational messaging and peer suggestions); and (2) "Coach Me" (tailored messaging to increase the intensity level of everyday activities and overcome barriers).
  Interventions: Other: Physical Activity (PA) Tracker App; Other: On Your Feet; Other: Coach Me
- PA App + On Your Feet + Proof Positive (Other): Participants in this arm will use a basic physical activity (PA) tracker app in conjunction with the following 2 features: (1) "On Your Feet" (sedentary activity monitoring with motivational messaging and peer suggestions); and (2) "Proof Positive" (explicit and implicit messaging to promote positive aging views).
  Interventions: Other: Physical Activity (PA) Tracker App; Other: On Your Feet; Other: Proof Positive
- PA App + On Your Feet (Other): Participants in this arm will use a basic physical activity (PA) tracker app in conjunction with the following feature: (1) "On Your Feet" (sedentary activity monitoring with motivational messaging and peer suggestions).
  Interventions: Other: Physical Activity (PA) Tracker App; Other: On Your Feet
- PA App + Coach Me + Proof Positive (Other): Participants in this arm will use a basic physical activity (PA) tracker app in conjunction with the following 2 features: (1) "Coach Me" (tailored messaging to increase the intensity level of everyday activities and overcome barriers); and (2) "Proof Positive" (explicit and implicit messaging to promote positive aging views).
  Interventions: Other: Physical Activity (PA) Tracker App; Other: Coach Me; Other: Proof Positive
- PA App + Coach Me (Other): Participants in this arm will use a basic physical activity (PA) tracker app in conjunction with the following feature: (1) "Coach Me" (tailored messaging to increase the intensity level of everyday activities and overcome barriers).
  Interventions: Other: Physical Activity (PA) Tracker App; Other: Coach Me
- PA App + Proof Positive (Other): Participants in this arm will use a basic physical activity (PA) tracker app in conjunction with the following feature: (1) "Proof Positive" (explicit and implicit messaging to promote positive aging views).
  Interventions: Other: Physical Activity (PA) Tracker App; Other: Proof Positive
- PA App (Other): Participants in this arm will use a basic physical activity (PA) tracker app without any additional features.
  Interventions: Other: Physical Activity (PA) Tracker App

INTERVENTIONS:
Other: Physical Activity (PA) Tracker App — This PA tracker app auto-monitors PA and provides a text-based summary of goal progress, thereby targeting self-regulation and outcome expectation.
Other: On Your Feet — On Your Feet is a specialty app feature designed to be paired with a PA tracker app and reduce sedentary activity-a health risk factor largely independent of insufficient PA. This feature utilizes self-regulatory and behavior change techniques including goal-setting, progress feedback, and prompting. Accumulated sedentary activity time is displayed alongside self-selected goals; reminders to stand are sent at a user-specified frequency; and general tips and previously compiled, older adult-identified strategies to reduce sedentary activity are texted. Additionally, messages about the benefits of reducing sedentary activity and overcoming barriers are sent.
  Arms: PA App + On Your Feet; PA App + On Your Feet + Coach Me; PA App + On Your Feet + Proof Positive; PA App+ On Your Feet+ CoachMe+ Proof Pos
Other: Coach Me — Coach Me is a specialty app feature designed to be paired with a PA tracker app and includes daily messages that assist older adults in discovering practical ways to integrate PA into their daily routines and overcoming PA barriers. Blending PA with productive activity facilitates PA engagement in older adults. In Coach Me, suggestions on how to intensify daily activities are tailored based on user selections from an activity inventory. This app feature helps older adults become more active in a minimally intrusive way, while allowing for engagement in productive and meaningful activities. Coach Me asks users to select obstacles to PA encountered in the previous week. Based on those selections, the app sends strategies on how to overcome those barriers, thereby targeting self-efficacy.
  Arms: PA App + Coach Me; PA App + Coach Me + Proof Positive; PA App + On Your Feet + Coach Me; PA App+ On Your Feet+ CoachMe+ Proof Pos
Other: Proof Positive — Proof Positive is a specialty app feature designed to be paired with a PA tracker app and capitalizes on the beneficial effects that exposure to positive aging messages and stereotypes has on health and PA. When activated, users (a) receive texts describing how old age does not equate to physical inability, (b) obtain information about the benefits of growing older, and (c) are presented with a weekly positive aging stereotype task modeled after a computerized series. This last function exposes users to blocks of "positive priming words." Primers are quickly flashed to allow perception without awareness while users focus on a simple icon that represents PA. Icons are intended to provide an additional PA cue, maintain user interest, and increase the external validity.
  Arms: PA App + Coach Me + Proof Positive; PA App + On Your Feet + Proof Positive; PA App + Proof Positive; PA App+ On Your Feet+ CoachMe+ Proof Pos

SUMMARY:
The purpose of this study is to develop, test, and optimize a physical activity (PA)-tracking smartphone app and specialty features, which are designed to facilitate older adults' PA by targeting common barriers in this population. For example, one feature sends messages throughout the day about the good things about growing older to combat negative views about aging which has been linked to decreased PA. Participants will include older adult smartphone users who are between the ages of 65 and 84 and are not very physically active. In phase one of the study, three groups of five older adults will be formed to test the PA-tracking app and one of three specialty features for a two-week period, followed by a focus group to learn about the older adults' experiences. In phase two, approximately 100 participants will be randomly assigned to one of eight groups that include various combinations of specialty features with the PA tracker, for the purpose of pilot testing the app for a four-month period. Testing will occur at the beginning and the end of the four-month intervention period, and will measure PA levels, sedentary activity time, self-reported PA, and functional mobility.

DETAILED DESCRIPTION:
In this study, we will optimize a set of tailored specialty app features designed to be paired with a physical activity (PA)-tracking app to boost older adults' PA. This package, termed the MovingUp suite, is distinct from generic fitness apps because it blends a set of specialized components that reflect empirically supported constructs from social cognitive and stereotype embodiment theory with evidence-based behavior change techniques (e.g., self-regulation) foundational to basic activity monitoring. Specialty features include: (a) explicit and implicit messaging to promote positive aging views; (b) sedentary activity monitoring with motivational messaging and peer suggestions; and (c) tailored messaging to increase the intensity level of everyday activities and overcome barriers. We will utilize a highly efficient, innovative methodological approach-Multiphase Optimization Strategy (MOST)-to provide an experimental context for evaluating the viability of each MovingUp specialty feature.

Aim 1: Assess the feasibility and acceptability of the three MovingUp specialty features. We will first examine MovingUp's feasibility and acceptability in three groups of five older adults (aged 65-84 years). A basic PA-tracking app plus one of three specialty features will be introduced-a different feature per group-at an orientation session. Groups will then test their assigned specialty feature with the PA tracker for two weeks. This step will involve real-time user data collection, check-ins via phone, and follow-up focus groups. Feasibility and acceptability will be determined by analyzing participants' usage patterns, evaluations of MovingUp features (based on a health technology usability scale and focus group interviews), and self-reported facilitators and barriers to successful app use. Our team will review the data and integrate changes as needed, producing an upgraded prototype to be assessed in Aim 2.

Aim 2: Conduct a pilot test to examine performance characteristics and PA-relevant outcomes of MovingUp's specialty features. Aim 2 includes the MOST Screening Phase: theory-guided experimentation to identify viable components within a multifaceted preliminary intervention plan. Using a factorial design as specified in MOST procedures, 100 underactive older adults (i.e., accumulating <150 minutes of moderate intensity activity per week) will be randomly assigned to one of eight conditions which reflect all possible combinations of presence vs. absence of the three respective specialty features, given usage of a PA tracker app. At the end of a four-month intervention period, for each specialty feature we will examine changes from baseline in PA-related outcomes including: objective PA (primary outcome), sedentary activity time, self-reported PA, and functional mobility. We will also examine the app components' relationships to theoretically postulated mediating constructs (self-efficacy, self-regulation, outcome expectation, social support, aging self-perception, and views of aging). In addition, we will document usage rate, sustained usage, and perceived usefulness for achieving PA goals for each suite component.

Aim 3: Synthesize information from Aim 2 to design an optimized MovingUp suite to be evaluated in a future RCT. Our study team will interpret and synthesize the array of resulting data to derive an optimized MovingUp suite. A set of pre-specified criteria will be used to guide selection of components in the optimized app. Using preliminary efficacy data, the stage will be set for a fully powered RCT of MovingUp's beneficial effects in comparison to alternate technologies such as web-based or mHealth solutions.

This project will help establish a methodological foundation for future attempts to enhance PA apps via the addition of theoretically based component features. Moreover, it will provide insights into the theoretical underpinnings of successful PA interventions for older adults, leading to information that transcends any single technology-based solution.

ELIGIBILITY:
Inclusion Criteria:

* 65-84 years old
* English speaking
* reside in Los Angeles
* score ≥5 on a 6-item cognitive screener
* report <150 minutes of moderate to vigorous PA/week as per a single-item screener
* ambulatory
* able to safely participate in physical activity as determined by the Revised Physical Activity Readiness Questionnaire (rPARQ) or proof of medical clearance from a physician
* smartphone owner for ≥3 months
* observed ability to reliably access and operate a smartphone during orientation.

Exclusion Criteria:

* ≥85 years old, based on limited smartphone ownership and to reduce sample variability

Ages: 65 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 111 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2021-01-12 (Actual); Study Completion 2021-01-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Front Porch Center for Innovation and Wellbeing, Glendale, California
  - University of Southern California, Los Angeles, California

IPD SHARING:
Plan to Share IPD: Yes
This proposal does not involve a multisite trial. The University of Southern California is the only project site. Funds greater than $500,000 are not requested and thus data-sharing is not required. The final results and dataset of the project, however, will be published and shared according to the NIH regulations in order to improve the transparency of the research.
Time Frame: Final results and dataset will be made available no later than the publication of the main findings from the final dataset. The data will remain in the repository indefinitely.
Access Criteria: Persons accessing the data through the repository must agree to certain terms of use to include the following: (1) must use data for research purposes only and not for investigation of specific research subjects; (2) must make no use of the identity of any research subject discovered inadvertently, and to advise the repository of any such discovery; (3) must agree not to redistribute data or other materials without the written agreement; and (4) must reference the recommended bibliographic citation in any publication that employs resources provided by the repository. Authors of publications based on shared data are required to send citations of their published works to the repository for inclusion in a database of related publications.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 197 screened for eligibility. 111 signed consent. 107 were randomized. 105 included in intent-to-treat analysis.
Pre-assignment Details: Two participants withdrew from the study after the study team randomized them but before the participants learned what group to which they were assigned. These two individuals were not included in the intent-to-treat analysis.
Groups:
- AT App+ On Your Feet+ CoachMe+ Proof Pos: Basic activity tracker (AT) app in conjunction with the following 3 features: (1) "On Your Feet" (sedentary activity monitoring with motivational messaging and peer suggestions); (2) "Coach Me" (tailored messaging to increase the intensity level of everyday activities and overcome barriers); and (3) "Proof Positive" (explicit and implicit messaging to promote positive aging views).
  AT App: app auto-monitors PA and provides a text-based summary of goal progress.
  On Your Feet: app feature designed reduce sedentary activity. Utilizes goal-setting, progress feedback, and prompting. Accumulated sedentary activity time is displayed alongside self-selected goals; reminders to stand are sent; and general tips and strategies to reduce sedentary activity and messages about the benefits of reducing sedentary activity and overcoming barriers are sent.
  Coach Me: app feature designed to assist older adults in discovering practical ways to integrate PA into their daily routines and overcoming PA barriers. Tailored suggestions on how to intensify daily activities and how to overcome barriers are sent.
  Proof Positive: app feature capitalizes on the beneficial effects exposure to positive aging messages and stereotypes has on health. Users receive texts describing how old age does not equate to physical inability, information about the benefits of growing older, and positive aging stereotype task.
- AT App + On Your Feet + Coach Me: Participants in this arm will use a basic activity tracker (AT) app in conjunction with the following 2 features: (1) "On Your Feet" (sedentary activity monitoring with motivational messaging and peer suggestions); and (2) "Coach Me" (tailored messaging to increase the intensity level of everyday activities and overcome barriers).
  AT App: app auto-monitors PA and provides a text-based summary of goal progress.
  On Your Feet: app feature designed reduce sedentary activity. Utilizes goal-setting, progress feedback, and prompting. Accumulated sedentary activity time is displayed alongside self-selected goals; reminders to stand are sent; and general tips and strategies to reduce sedentary activity and messages about the benefits of reducing sedentary activity and overcoming barriers are sent.
  Coach Me: app feature designed to assist older adults in discovering practical ways to integrate PA into their daily routines and overcoming PA barriers. Tailored suggestions on how to intensify daily activities and how to overcome barriers are sent.
- AT App + On Your Feet + Proof Positive: Participants in this arm will use a basic activity tracker (AT) app in conjunction with the following 2 features: (1) "On Your Feet" (sedentary activity monitoring with motivational messaging and peer suggestions); and (2) "Proof Positive" (explicit and implicit messaging to promote positive aging views).
  AT App: app auto-monitors physical activity and provides a text-based summary of goal progress.
  On Your Feet: app feature designed reduce sedentary activity. Utilizes goal-setting, progress feedback, and prompting. Accumulated sedentary activity time is displayed alongside self-selected goals; reminders to stand are sent; and general tips and strategies to reduce sedentary activity and messages about the benefits of reducing sedentary activity and overcoming barriers are sent.
  Proof Positive: app feature capitalizes on the beneficial effects exposure to positive aging messages and stereotypes has on health. Users receive texts describing how old age does not equate to physical inability, information about the benefits of growing older, and positive aging stereotype task.
- AT App + On Your Feet: Participants in this arm will use a basic activity tracker (AT) app in conjunction with the following feature: (1) "On Your Feet" (sedentary activity monitoring with motivational messaging and peer suggestions).
  AT App: app auto-monitors physical activity and provides a text-based summary of goal progress.
  On Your Feet: app feature designed reduce sedentary activity. Utilizes goal-setting, progress feedback, and prompting. Accumulated sedentary activity time is displayed alongside self-selected goals; reminders to stand are sent; and general tips and strategies to reduce sedentary activity and messages about the benefits of reducing sedentary activity and overcoming barriers are sent.
- AT App + Coach Me + Proof Positive: Participants in this arm will use a basic activity tracker (AT) app in conjunction with the following 2 features: (1) "Coach Me" (tailored messaging to increase the intensity level of everyday activities and overcome barriers); and (2) "Proof Positive" (explicit and implicit messaging to promote positive aging views).
  AT App: This physical activity tracker app auto-monitors physical activity and provides a text-based summary of goal progress, thereby targeting self-regulation and outcome expectation.
  Coach Me: app feature designed to assist older adults in discovering practical ways to integrate PA into their daily routines and overcoming PA barriers. Tailored suggestions on how to intensify daily activities and how to overcome barriers are sent.
  Proof Positive: app feature capitalizes on the beneficial effects exposure to positive aging messages and stereotypes has on health. Users receive texts describing how old age does not equate to physical inability, information about the benefits of growing older, and positive aging stereotype task.
- AT App + Coach Me: Participants in this arm will use a basic activity tracker (AT) app in conjunction with the following feature: (1) "Coach Me" (tailored messaging to increase the intensity level of everyday activities and overcome barriers).
  AT App: This physical activity tracker app auto-monitors physical activity and provides a text-based summary of goal progress, thereby targeting self-regulation and outcome expectation.
  Coach Me: app feature designed to assist older adults in discovering practical ways to integrate PA into their daily routines and overcoming PA barriers. Tailored suggestions on how to intensify daily activities and how to overcome barriers are sent.
- AT App + Proof Positive: Participants in this arm will use a basic activity tracker (AT) app in conjunction with the following feature: (1) "Proof Positive" (explicit and implicit messaging to promote positive aging views).
  AT App: This physical activity tracker app auto-monitors physical activity and provides a text-based summary of goal progress, thereby targeting self-regulation and outcome expectation.
  Proof Positive: app feature capitalizes on the beneficial effects exposure to positive aging messages and stereotypes has on health. Users receive texts describing how old age does not equate to physical inability, information about the benefits of growing older, and positive aging stereotype task.
- AT App: Participants in this arm will use a basic physical activity (PA) tracker app without any additional features.
  AT App: This physical activity tracker app auto-monitors physical activity and provides a text-based summary of goal progress, thereby targeting self-regulation and outcome expectation.
Period: Overall Study
Arm/Group | AT App+ On Your Feet+ CoachMe+ Proof Pos | AT App + On Your Feet + Coach Me | AT App + On Your Feet + Proof Positive | AT App + On Your Feet | AT App + Coach Me + Proof Positive | AT App + Coach Me | AT App + Proof Positive | AT App
Started | 13 | 13 | 14 | 14 | 14 | 12 | 15 | 12
Non-completer But Included in ITT | 1 | 1 | 1 | 1 | 2 | 0 | 0 | 1
Non-completer But NOT Included in ITT | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Completed | 11 | 12 | 12 | 13 | 12 | 12 | 15 | 11
Not Completed | 2 | 1 | 2 | 1 | 2 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 2 | 1 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- AT App + On Your Feet+ CoachMe+ Proof Pos: Basic physical activity tracker (AT) app in conjunction with the following 3 features: (1) "On Your Feet" (sedentary activity monitoring with motivational messaging and peer suggestions); (2) "Coach Me" (tailored messaging to increase the intensity level of everyday activities and overcome barriers); and (3) "Proof Positive" (explicit and implicit messaging to promote positive aging views).
  Activity Tracker App: app auto-monitors physical activity and provides a text-based summary of goal progress.
  On Your Feet: app feature designed reduce sedentary activity. Utilizes goal-setting, progress feedback, and prompting. Accumulated sedentary activity time is displayed alongside self-selected goals; reminders to stand are sent; and general tips and strategies to reduce sedentary activity and messages about the benefits of reducing sedentary activity and overcoming barriers are sent.
  Coach Me: app feature designed to assist older adults in discovering practical ways to integrate PA into their daily routines and overcoming PA barriers. Tailored suggestions on how to intensify daily activities and how to overcome barriers are sent.
  Proof Positive: app feature capitalizes on the beneficial effects exposure to positive aging messages and stereotypes has on health. Users receive texts describing how old age does not equate to physical inability, information about the benefits of growing older, and positive aging stereotype task.
- AT App + On Your Feet + Coach Me: Participants in this arm will use a basic physical activity tracker (AT) app in conjunction with the following 2 features: (1) "On Your Feet" (sedentary activity monitoring with motivational messaging and peer suggestions); and (2) "Coach Me" (tailored messaging to increase the intensity level of everyday activities and overcome barriers).
  Activity Tracker App: app auto-monitors physical activity and provides a text-based summary of goal progress.
  On Your Feet: app feature designed reduce sedentary activity. Utilizes goal-setting, progress feedback, and prompting. Accumulated sedentary activity time is displayed alongside self-selected goals; reminders to stand are sent; and general tips and strategies to reduce sedentary activity and messages about the benefits of reducing sedentary activity and overcoming barriers are sent.
  Coach Me: app feature designed to assist older adults in discovering practical ways to integrate PA into their daily routines and overcoming PA barriers. Tailored suggestions on how to intensify daily activities and how to overcome barriers are sent.
- AT App + On Your Feet + Proof Positive: Participants in this arm will use a basic physical activity tracker (AT) app in conjunction with the following 2 features: (1) "On Your Feet" (sedentary activity monitoring with motivational messaging and peer suggestions); and (2) "Proof Positive" (explicit and implicit messaging to promote positive aging views).
  Activity Tracker App: app auto-monitors physical activity and provides a text-based summary of goal progress.
  On Your Feet: app feature designed reduce sedentary activity. Utilizes goal-setting, progress feedback, and prompting. Accumulated sedentary activity time is displayed alongside self-selected goals; reminders to stand are sent; and general tips and strategies to reduce sedentary activity and messages about the benefits of reducing sedentary activity and overcoming barriers are sent.
  Proof Positive: app feature capitalizes on the beneficial effects exposure to positive aging messages and stereotypes has on health. Users receive texts describing how old age does not equate to physical inability, information about the benefits of growing older, and positive aging stereotype task.
- AT App + On Your Feet: Participants in this arm will use a basic physical activity tracker (AT) app in conjunction with the following feature: (1) "On Your Feet" (sedentary activity monitoring with motivational messaging and peer suggestions).
  Activity Tracker App: app auto-monitors physical activity and provides a text-based summary of goal progress.
  On Your Feet: app feature designed reduce sedentary activity. Utilizes goal-setting, progress feedback, and prompting. Accumulated sedentary activity time is displayed alongside self-selected goals; reminders to stand are sent; and general tips and strategies to reduce sedentary activity and messages about the benefits of reducing sedentary activity and overcoming barriers are sent.
- AT App + Coach Me + Proof Positive: Participants in this arm will use a basic physical activity tracker (AT) app in conjunction with the following 2 features: (1) "Coach Me" (tailored messaging to increase the intensity level of everyday activities and overcome barriers); and (2) "Proof Positive" (explicit and implicit messaging to promote positive aging views).
  Activity Tracker App: app auto-monitors physical activity and provides a text-based summary of goal progress, thereby targeting self-regulation and outcome expectation.
  Coach Me: app feature designed to assist older adults in discovering practical ways to integrate PA into their daily routines and overcoming PA barriers. Tailored suggestions on how to intensify daily activities and how to overcome barriers are sent.
  Proof Positive: app feature capitalizes on the beneficial effects exposure to positive aging messages and stereotypes has on health. Users receive texts describing how old age does not equate to physical inability, information about the benefits of growing older, and positive aging stereotype task.
- AT App + Coach Me: Participants in this arm will use a basic physical activity tracker (AT) app in conjunction with the following feature: (1) "Coach Me" (tailored messaging to increase the intensity level of everyday activities and overcome barriers).
  Activity Tracker App: app auto-monitors physical activity and provides a text-based summary of goal progress, thereby targeting self-regulation and outcome expectation.
  Coach Me: app feature designed to assist older adults in discovering practical ways to integrate PA into their daily routines and overcoming PA barriers. Tailored suggestions on how to intensify daily activities and how to overcome barriers are sent.
- AT App + Proof Positive: Participants in this arm will use a basic physical activity tracker (AT) app in conjunction with the following feature: (1) "Proof Positive" (explicit and implicit messaging to promote positive aging views).
  Activity Tracker App: app auto-monitors physical activity and provides a text-based summary of goal progress, thereby targeting self-regulation and outcome expectation.
  Proof Positive: app feature capitalizes on the beneficial effects exposure to positive aging messages and stereotypes has on health. Users receive texts describing how old age does not equate to physical inability, information about the benefits of growing older, and positive aging stereotype task.
- AT App: Participants in this arm will use a basic physical activity tracker (AT) app without any additional features.
  Activity Tracker App: app auto-monitors physical activity and provides a text-based summary of goal progress, thereby targeting self-regulation and outcome expectation.
- Total: Total of all reporting groups
Arm/Group | AT App + On Your Feet+ CoachMe+ Proof Pos | AT App + On Your Feet + Coach Me | AT App + On Your Feet + Proof Positive | AT App + On Your Feet | AT App + Coach Me + Proof Positive | AT App + Coach Me | AT App + Proof Positive | AT App | Total
Number analyzed (Participants) | 12 | 13 | 13 | 14 | 14 | 12 | 15 | 12 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.4 (5.3) | 72.1 (4.2) | 71.6 (3.4) | 72.7 (4.6) | 71.5 (4.3) | 72.2 (4.2) | 72.4 (4.2) | 74.4 (6.4) | 72.2 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 10 | 8 | 9 | 11 | 12 | 11 | 77
  Male | 4 | 5 | 3 | 6 | 5 | 1 | 3 | 1 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 5
  Not Hispanic or Latino | 11 | 13 | 11 | 14 | 13 | 12 | 15 | 9 | 98
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 1 | 4 | 3 | 0 | 1 | 1 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 4 | 4 | 4 | 1 | 3 | 5 | 3 | 28
  White | 7 | 7 | 8 | 6 | 10 | 9 | 9 | 8 | 64
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 13 | 13 | 14 | 14 | 12 | 15 | 12 | 105
Education [Count of Participants; unit: Participants] — Participant's reported level of education dichotomized into "high school or some college/trade school" or "college graduate"
  Participants
    High school or some college/trade school | 3 | 7 | 2 | 1 | 3 | 1 | 4 | 4 | 25
    College graduate | 9 | 6 | 11 | 13 | 11 | 11 | 11 | 8 | 80
Self-rated smartphone ability [Mean (Standard Deviation); unit: units on a scale] — Asked participants to "rate your ability to use your smartphone" on a scale: 1=poor to 10=excellent.
  units on a scale | 7.6 (1.8) | 7.2 (2.7) | 7.2 (1.3) | 7.1 (1.4) | 7.8 (2.1) | 6.5 (1.5) | 7.0 (2.1) | 6.3 (2.1) | 7.1 (1.9)
Health Conditions [Count of Participants; unit: Participants] — Only health conditions reported by 10 or more participants are included.
  Participants
    Arthritis | 3 | 2 | 7 | 7 | 3 | 5 | 8 | 3 | 38
    Cancer | 1 | 4 | 2 | 1 | 4 | 5 | 3 | 3 | 23
    Depression | 1 | 3 | 3 | 2 | 0 | 4 | 4 | 2 | 19
    High blood pressure | 6 | 6 | 7 | 7 | 4 | 4 | 4 | 5 | 43
    High cholesterol | 6 | 7 | 8 | 6 | 4 | 5 | 4 | 5 | 45
    Diabetes | 1 | 3 | 2 | 1 | 3 | 3 | 0 | 1 | 14

OUTCOME MEASURES:

1. Primary Outcome: Daily Steps Change From Baseline to Month 4; Main Effect, and 2- and 3-way Interactions
Description: Step counts (objective physical activity) were measured using the activPAL thigh-worn accelerometer during a 72-hour monitoring period.
  Estimated average change is computed as the change in activPAL-tracked mean daily steps at Month 4 relative to baseline; this outcome is analyzed in a linear regression analysis model. All randomized participants who started the intervention and had valid activity monitor data were utilized in the model (ITT analysis)
Time Frame: 72-hour monitoring periods at Month 4 relative to baseline
Population: ITT population: all randomized participants who started the intervention and who had at least one valid activity monitoring period. Participants included underactive older adults who own a smartphone. Change in physical activity patterns of these individuals was measured.
Measure: Mean (Standard Deviation); unit: Average change in steps per day
Groups:
- Proof Positive On: All participants either received Proof Positive app feature (ON) or did not (OFF). This group represents all those who had the Proof Positive feature ON, regardless of what other features they may have also received, and also valid activity monitor data.
- Proof Positive Off: All participants either received Proof Positive app feature (ON) or did not (OFF). This group represents all those whose Proof Positive feature was OFF, regardless of what other features they may have also received, and also had valid activity monitor data.
- Coach Me On: All participants either received Coach Me app feature (ON) or did not (OFF). This group represents all those who had the Coach Me feature ON, regardless of what other features they may have also received, and also had valid activity monitor data.
- Coach Me Off: All participants either received Coach Me app feature (ON) or did not (OFF). This group represents all those whose Coach Me feature was OFF, regardless of what other features they may have also received, and also had valid activity monitor data.
- On Your Feet On: All participants either received On Your Feet app feature (ON) or did not (OFF). This group represents all those who had the On Your Feet feature ON, regardless of what other features they may have also received, and also had valid activity monitor data.
- On Your Feet Off: All participants either received On Your Feet app feature (ON) or did not (OFF). This group represents all those whose On Your Feet feature was OFF, regardless of what other features they may have also received, and also had valid activity monitor data.
Arm/Group | Proof Positive On | Proof Positive Off | Coach Me On | Coach Me Off | On Your Feet On | On Your Feet Off
Number analyzed (Participants) | 49 | 47 | 46 | 50 | 48 | 48
Average change in steps per day | -343.5 (2689.5) | -324.5 (2263.1) | -859.9 (2588.6) | 149.5 (2289.6) | -424.8 (2101.2) | -243.5 (2822.8)
Statistical Analysis 1: Comparison: Proof Positive On; The original mixed effects regression model effects consisted of three treatment main effects, three two-way treatment interactions, and one three-way treatment interaction. Values are unadjusted; Test type: Superiority; p = .37, Mixed Models Analysis — A single model was run including variables indicating Proof Positive (yes/no), Coach Me (yes/no), and On Your Feet (yes/no) and their interaction terms; Estimated mean change = -898.0, 95% CI 2-sided [-2884.82 to 1088.82]
Statistical Analysis 2: Comparison: Coach Me On; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .02, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Estimated mean change = -2602.1, 95% CI 2-sided [-4687.44 to -516.69]
Statistical Analysis 3: Comparison: On Your Feet On; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .23, Mixed Models Analysis; Estimated mean change = -1244.9, 95% CI 2-sided [-3287.60 to 797.85]
Statistical Analysis 4: Comparison: Proof Positive On vs Coach Me On; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.31, Mixed Models Analysis; Estimated mean change = 1468.5, 95% CI 2-sided [-1368.93 to 4306.02]
Statistical Analysis 5: Comparison: Proof Positive On vs On Your Feet On; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.78, Mixed Models Analysis; Estimated mean change = 388.1, 95% CI 2-sided [-2397.51 to 3173.62]
Statistical Analysis 6: Comparison: Coach Me On vs On Your Feet On; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.17, Mixed Models Analysis; Estimated mean change = 1991.2, 95% CI 2-sided [-865.52 to 4847.86]
Statistical Analysis 7: Comparison: Proof Positive On vs Coach Me On vs On Your Feet On; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.77, Mixed Models Analysis; Estimated mean change = -590.7, 95% CI 2-sided [-4591.17 to 3409.75]

2. Secondary Outcome: Daily Sitting Time (activPAL) Change From Baseline to Month 4
Description: Objective sedentary activity time was measured using the activPAL thigh-worn accelerometer during a 72-hour monitoring period. Expressed as average minutes/day.
Time Frame: 72-hour monitoring periods at Month 4 relative to baseline
Population: ITT population: all randomized participants who started the intervention and who had valid activity monitoring periods at baseline and post-test. Participants included underactive older adults who own a smartphone. Change in physical activity patterns of these individuals was measured.
Measure: Mean (Standard Deviation); unit: Change in minutes/day
Groups:
- Proof Positive On; Proof Positive Off: All participants either received Proof Positive app feature (on) or did not (off). The group includes participants who received combinations of the other two app feature interventions (Coach Me or No Coach Me; On Your Feet or No On Your Feet). The Proof Positive ITT group consists of 54 participants (approximately half of the total study sample) and is compared to a corresponding No Proof Positive group consisting of 51 participants (approximately half of the total study sample) in a main effect (Proof Positive versus No Proof Positive) statistical comparison.
- Coach Me On; Coach Me Off: All participants either received Coach Me app feature (on) or did not (off). The group includes participants who received combinations of the other two app feature interventions (Proof Positive or No Proof Positive; On Your Feet or No On Your Feet). The Coach Me ITT group consists of 51 participants (approximately half of the total study sample) and is compared to a corresponding No Coach Me group consisting of 54 participants (approximately half of the total study sample) in a main effect (Coach Me versus No Coach Me) statistical comparison.
- On Your Feet On; On Your Feet Off: All participants either received On Your Feet app feature (on) or did not (off). The group includes participants who received combinations of the other two app feature interventions (Coach Me or No Coach Me; Proof Positive or No Proof Positive). The On Your Feet ITT group consists of 52 participants (approximately half of the total study sample) and is compared to a corresponding No On Your Feet group consisting of 53 participants (approximately half of the total study sample) in a main effect (On Your Feet versus No On Your Feet) statistical comparison.
Arm/Group | Proof Positive On | Proof Positive Off | Coach Me On | Coach Me Off | On Your Feet On | On Your Feet Off
Number analyzed (Participants) | 49 | 47 | 46 | 50 | 48 | 48
Change in minutes/day | -11.6 (108.1) | 11.4 (128.9) | 19.3 (123.6) | -18.4 (112.2) | 25.7 (117.3) | -26.3 (115.5)
Statistical Analysis 1: Comparison: Proof Positive On vs Proof Positive Off; Test type: Superiority; p = 0.17, t-test, 1 sided — a priori threshold for statistical significance=0.1 for 1-sided t-test; no adjustments for multiple comparisons made; if the outcome is not in the hypothesized direction, values that meet or exceed the 0.1 threshold will not be considered significant; Mean Difference (Net) = -23, 90% CI 1-sided [upper limit 8.3], Standard Deviation 118.7
Statistical Analysis 2: Comparison: Coach Me On vs Coach Me Off; Test type: Superiority; p = 0.94, t-test, 1 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 37.7, 90% CI 1-sided [upper limit 68.8], Standard Deviation 117.8
Statistical Analysis 3: Comparison: On Your Feet On vs On Your Feet Off; Test type: Superiority; p = 0.99, t-test, 1 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 52.0, 90% CI 1-sided [upper limit 82.7], Standard Deviation 116.4

3. Secondary Outcome: Self-reported Physical Activity (PASE) Change From Baseline to Month 4
Description: Self-reported physical activity will be measured via the Physical Activity Scale for the Elderly (PASE). PASE is a ten-item instrument designed to assess engagement in physical activities commonly pursued by older adults, including those related to leisure, household, and occupational tasks. The tool is a valid and reliable measure of physical activity engagement in the older adult population. Scores range from 0 to 361. Higher scores indicate a higher level of activity.
Time Frame: baseline and 4 months
Population: ITT population: all randomized participants who started the intervention and who had valid questionnaire data at baseline and post-test. Participants included underactive older adults who own a smartphone. Change in physical activity patterns of these individuals was measured.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Proof Positive On | Proof Positive Off | Coach Me On | Coach Me Off | On Your Feet On | On Your Feet Off
Number analyzed (Participants) | 50 | 48 | 47 | 51 | 48 | 50
score on a scale | 4.0 (41.6) | 3.2 (59.3) | 6.2 (44.2) | 1.2 (56.5) | 5.6 (54.4) | 1.7 (47.5)
Statistical Analysis 1: Comparison: Proof Positive On vs Proof Positive Off; Test type: Superiority; p = 0.47, t-test, 1 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = .8, 90% CI 1-sided [lower limit -12.5], Standard Deviation 51
Statistical Analysis 2: Comparison: Coach Me On vs Coach Me Off; Test type: Superiority; p = 0.315, t-test, 1 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 5, 90% CI 1-sided [lower limit -8.3], Standard Deviation 51
Statistical Analysis 3: Comparison: On Your Feet On vs On Your Feet Off; Test type: Superiority; p = 0.355, t-test, 1 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 3.9, 90% CI 1-sided [lower limit -9.4], Standard Deviation 51

4. Secondary Outcome: Gait Speed (4-m Walk Test) Change From Baseline to Month 4
Description: Functional mobility will be assessed through a four-meter walk test, a commonly used, validated measure of physical and functional performance in older adults.
Time Frame: baseline and 4 months
Population: ITT population: all randomized participants who started the intervention and who had walk test data at baseline and post-test. Participants included underactive older adults who own a smartphone. Change was measured. Note: very few data were available due to COVID-19 restrictions negating continuation of data collection for this variable.
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | Proof Positive On | Proof Positive Off | Coach Me On | Coach Me Off | On Your Feet On | On Your Feet Off
Number analyzed (Participants) | 5 | 8 | 5 | 8 | 4 | 9
meters/second | -0.7 (0.9) | -0.1 (1.0) | -0.2 (1.2) | -0.4 (0.9) | -0.5 (1.0) | -0.2 (1.0)
Statistical Analysis 1: Comparison: Proof Positive On vs Proof Positive Off; Test type: Superiority; p = 0.86, t-test, 1 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -.6, 90% CI 1-sided [lower limit -1.3], Standard Deviation 1.0
Statistical Analysis 2: Comparison: Coach Me On vs Coach Me Off; Test type: Superiority; p = 0.38, t-test, 1 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = .2, 90% CI 1-sided [lower limit -0.6], Standard Deviation 1.0
Statistical Analysis 3: Comparison: On Your Feet On vs On Your Feet Off; Test type: Superiority; p = 0.66, t-test, 1 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -.3, 90% CI 1-sided [lower limit -1.1], Standard Deviation 1.0

5. Secondary Outcome: Self-efficacy for Physical Activity (Health Beliefs Survey) Change From Baseline
Description: The potential mediators of physical activity self-efficacy, self-regulation, outcome expectation, and social support will each be measured separately using subscales of the 78-item physical activity portion of the Health Beliefs Survey. Subscales demonstrate sufficient internal consistencies (Cronbach's α=0.68-0.90) and are predictive of physical activity. Higher scores indicate greater self-efficacy. Possible scores for the self-efficacy subscale range from 0-100.
Time Frame: baseline and 4 months
Population: ITT population: all randomized participants who started the intervention and who had valid questionnaire data at baseline and post-test. Participants included underactive older adults who own a smartphone. Change was measured.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Proof Positive On | Proof Positive Off | Coach Me On | Coach Me Off | On Your Feet On | On Your Feet Off
Number analyzed (Participants) | 50 | 48 | 47 | 51 | 48 | 50
units on a scale | -4.8 (18.5) | -2.9 (19.8) | -4.4 (17.4) | -3.4 (20.7) | -1.4 (16.7) | -6.2 (21)
Statistical Analysis 1: Comparison: Proof Positive On vs Proof Positive Off; Test type: Superiority; p = 0.69, t-test, 1 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -1.9, 90% CI 1-sided [lower limit -6.9], Standard Deviation 19.2
Statistical Analysis 2: Comparison: Coach Me On vs Coach Me Off; Test type: Superiority; p = 0.60, t-test, 1 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -1.0, 90% CI 1-sided [lower limit -6.0], Standard Deviation 19.2
Statistical Analysis 3: Comparison: On Your Feet On vs On Your Feet Off; Test type: Superiority; p = 0.11, t-test, 1 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 4.8, 90% CI 1-sided [lower limit -0.2], Standard Deviation 19.0

6. Secondary Outcome: Self-regulation of Physical Activity (Health Beliefs Survey Physical Activity Portion) Change From Baseline
Description: The potential mediators of physical activity self-efficacy, self-regulation, outcome expectation, and social support will each be measured separately using subscales of the 78-item physical activity portion of the Health Beliefs Survey. Subscales demonstrate sufficient internal consistencies (Cronbach's α=0.68-0.90) and are predictive of physical activity. Higher scores indicate greater self-regulation behaviors. Possible scores for the self-regulation subscale range from 1-5.
Time Frame: baseline and 4 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Proof Positive On | Proof Positive Off | Coach Me On | Coach Me Off | On Your Feet On | On Your Feet Off
Number analyzed (Participants) | 50 | 48 | 47 | 51 | 48 | 50
score on a scale | 0.8 (1.0) | 1.2 (1.0) | 0.9 (1.0) | 1.0 (1.1) | 1.1 (1.2) | 0.9 (0.9)
Statistical Analysis 1: Comparison: Proof Positive On vs Proof Positive Off; Test type: Superiority; p = 0.94, t-test, 1 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.4, 90% CI 1-sided [lower limit -0.7], Standard Deviation 1.0
Statistical Analysis 2: Comparison: Coach Me On vs Coach Me Off; Test type: Superiority; p = 0.73, t-test, 1 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.1, 90% CI 1-sided [lower limit -0.4], Standard Deviation 1.1
Statistical Analysis 3: Comparison: On Your Feet On vs On Your Feet Off; Test type: Superiority; p = 0.22, t-test, 1 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.2, 90% CI 1-sided [lower limit -0.1], Standard Deviation 1.1

7. Secondary Outcome: Family Social Support for Physical Activity (Health Beliefs Survey Physical Activity Portion) Change From Baseline
Description: The potential mediators of physical activity self-efficacy, self-regulation, outcome expectation, and social support will each be measured separately using subscales of the 78-item physical activity portion of the Health Beliefs Survey. Subscales demonstrate sufficient internal consistencies (Cronbach's α=0.68-0.90) and are predictive of physical activity. Higher scores indicate greater family social support for physical activity. Possible scores for the family social support subscale range from 1 - 5.
Time Frame: baseline and 4 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Proof Positive On | Proof Positive Off | Coach Me On | Coach Me Off | On Your Feet On | On Your Feet Off
Number analyzed (Participants) | 47 | 47 | 45 | 49 | 46 | 48
score on a scale | 0.2 (1.2) | 0.2 (1.3) | -0.0 (1.1) | 0.4 (1.3) | 0.2 (1.1) | 0.2 (1.4)
Statistical Analysis 1: Comparison: Proof Positive On vs Proof Positive Off; Test type: Superiority; p = 0.46, t-test, 1 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.0, 90% CI 1-sided [lower limit -0.3], Standard Deviation 1.3
Statistical Analysis 2: Comparison: Coach Me On vs Coach Me Off; Test type: Superiority; p = 0.96, t-test, 1 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.4, 90% CI 1-sided [lower limit -0.7], Standard Deviation 1.2
Statistical Analysis 3: Comparison: On Your Feet On vs On Your Feet Off; Test type: Superiority; p = 0.495, t-test, 1 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.0, 90% CI 1-sided [lower limit -0.3], Standard Deviation 1.3

8. Secondary Outcome: Outcome Expectation for Physical Activity (Health Beliefs Survey Physical Activity Portion) Change From Baseline
Description: The potential mediators of physical activity self-efficacy, self-regulation, outcome expectation, and social support will each be measured separately using subscales of the 78-item physical activity portion of the Health Beliefs Survey. Subscales demonstrate sufficient internal consistencies (Cronbach's α=0.68-0.90) and are predictive of physical activity. Higher scores indicate greater outcome expectations. Possible scores for the outcome expectation subscale range from 1-25
Time Frame: baseline and 4 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Proof Positive On | Proof Positive Off | Coach Me On | Coach Me Off | On Your Feet On | On Your Feet Off
Number analyzed (Participants) | 47 | 47 | 46 | 48 | 46 | 48
score on a scale | -0.4 (4.2) | -0.5 (4.8) | -1.1 (4.0) | 0.2 (4.8) | -0.1 (3.8) | -0.8 (5.0)
Statistical Analysis 1: Comparison: Proof Positive On vs Proof Positive Off; Test type: Superiority; p = 0.445, t-test, 1 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.1, 90% CI 1-sided [lower limit -1.1], Standard Deviation 4.5
Statistical Analysis 2: Comparison: Coach Me On vs Coach Me Off; Test type: Superiority; p = 0.92, t-test, 1 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -1.3, 90% CI 1-sided [lower limit -2.5], Standard Deviation 4.4
Statistical Analysis 3: Comparison: On Your Feet On vs On Your Feet Off; Test type: Superiority; p = 0.23, t-test, 1 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.7, 90% CI 1-sided [lower limit -0.5], Standard Deviation 4.5

9. Secondary Outcome: Aging Self-perceptions (Attitudes Toward Own Aging) Change From Baseline
Description: Aging self-perceptions will be assessed by the Attitudes Toward Own Aging subscale of the Philadelphia Geriatrics Center Morale Scale. This five-question tool captures the subjective aging experience, shows moderate internal consistency (Cronbach's α=0.61-0.64), and predicts mortality risk. Scores can range from 0 to 5. A higher score indicates more positive aging self-perceptions.
Time Frame: baseline and 4 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Proof Positive On | Proof Positive Off | Coach Me On | Coach Me Off | On Your Feet On | On Your Feet Off
Number analyzed (Participants) | 50 | 48 | 47 | 51 | 48 | 50
score on a scale | 0.2 (1.1) | 0.4 (1.1) | 0.1 (0.9) | 0.5 (1.3) | 0.4 (1.2) | 0.2 (1.0)
Statistical Analysis 1: Comparison: Proof Positive On vs Proof Positive Off; Test type: Superiority; p = 0.78, t-test, 1 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.2, 90% CI 1-sided [lower limit -0.5], Standard Deviation 1.1
Statistical Analysis 2: Comparison: Coach Me On vs Coach Me Off; Test type: Superiority; p = 0.98, t-test, 1 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.4, 90% CI 1-sided [lower limit -0.7], Standard Deviation 1.1
Statistical Analysis 3: Comparison: On Your Feet On vs On Your Feet Off; Test type: Superiority; p = 0.13, t-test, 1 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.2, 90% CI 1-sided [lower limit -0.1], Standard Deviation 1.1

10. Secondary Outcome: Views of Aging--Psychosocial Loss (Attitudes to Ageing Questionnaire) Change From Baseline
Description: Views of aging will be measured using the Attitudes to Ageing Questionnaire. This 24-item assessment identifies subjective views about age-related changes in multiple domains, is cross-culturally valid, and is psychometrically sound (Cronbach's α=0.68-0.84). Its subscales include psychosocial loss, physical change, and psychological growth. A higher score for psychosocial loss indicates more negative attitude (min 8; max 40).
Time Frame: baseline and 4 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Proof Positive On | Proof Positive Off | Coach Me On | Coach Me Off | On Your Feet On | On Your Feet Off
Number analyzed (Participants) | 50 | 47 | 47 | 50 | 47 | 50
score on a scale | -0.6 (3.8) | -0.1 (4.8) | -0.3 (5.0) | -0.3 (3.6) | 0.3 (4.0) | -0.9 (4.5)
Statistical Analysis 1: Comparison: Proof Positive On vs Proof Positive Off; Test type: Superiority; p = 0.285, t-test, 1 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.5, 90% CI 1-sided [upper limit 0.6], Standard Deviation 4.3
Statistical Analysis 2: Comparison: Coach Me On vs Coach Me Off; Test type: Superiority; p = 0.50, t-test, 1 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.0, 90% CI 1-sided [upper limit 1.1], Standard Deviation 4.3
Statistical Analysis 3: Comparison: On Your Feet On vs On Your Feet Off; Test type: Superiority; p = 0.92, t-test, 1 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 1.2, 90% CI 1-sided [upper limit 2.3], Standard Deviation 4.3

11. Secondary Outcome: Views of Aging--Physical Change (Attitudes to Ageing Questionnaire) Change From Baseline
Description: Views of aging will be measured using the Attitudes to Ageing Questionnaire. This 24-item assessment identifies subjective views about age-related changes in multiple domains, is cross-culturally valid, and is psychometrically sound (Cronbach's α=0.68-0.84). Its subscales include psychosocial loss, physical change, and psychological growth. A higher score on physical change indicates more positive attitude (min 8; max 40)
Time Frame: baseline and 4 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Proof Positive On | Proof Positive Off | Coach Me On | Coach Me Off | On Your Feet On | On Your Feet Off
Number analyzed (Participants) | 48 | 45 | 45 | 48 | 46 | 47
score on a scale | 0.6 (4.2) | 0.4 (4.1) | 0.1 (3.2) | 0.9 (4.9) | 0.5 (4.6) | 0.6 (3.7)
Statistical Analysis 1: Comparison: Proof Positive On vs Proof Positive Off; Test type: Superiority; p = 0.42, t-test, 1 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.2, 90% CI 1-sided [lower limit -0.9], Standard Deviation 4.2
Statistical Analysis 2: Comparison: Coach Me On vs Coach Me Off; Test type: Superiority; p = 0.82, t-test, 1 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.8, 90% CI 1-sided [lower limit -1.9], Standard Deviation 4.2
Statistical Analysis 3: Comparison: On Your Feet On vs On Your Feet Off; Test type: Superiority; p = 0.58, t-test, 1 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.1, 90% CI 1-sided [lower limit -1.2], Standard Deviation 4.2

12. Secondary Outcome: Views of Aging--Psychological Growth (Attitudes to Ageing Questionnaire) Change From Baseline
Description: Views of aging will be measured using the Attitudes to Ageing Questionnaire. This 24-item assessment identifies subjective views about age-related changes in multiple domains, is cross-culturally valid, and is psychometrically sound (Cronbach's α=0.68-0.84). Its subscales include psychosocial loss, physical change, and psychological growth. A higher score on psychological growth indicates more positive attitude (min 8; max 40).
Time Frame: baseline and 4 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Proof Positive On | Proof Positive Off | Coach Me On | Coach Me Off | On Your Feet On | On Your Feet Off
Number analyzed (Participants) | 48 | 48 | 45 | 51 | 48 | 48
score on a scale | 0.0 (4.0) | -0.1 (3.9) | -0.0 (3.7) | -0.0 (4.1) | -0.1 (4.1) | 0.1 (3.7)
Statistical Analysis 1: Comparison: Proof Positive On vs Proof Positive Off; Test type: Superiority; p = 0.45, t-test, 1 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.1, 90% CI 1-sided [lower limit -0.9], Standard Deviation 4.0
Statistical Analysis 2: Comparison: Coach Me On vs Coach Me Off; Test type: Superiority; p = 0.49, t-test, 1 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.0, 90% CI 1-sided [lower limit -1.0], Standard Deviation 3.9
Statistical Analysis 3: Comparison: On Your Feet On vs On Your Feet Off; Test type: Superiority; p = 0.61, t-test, 1 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.2, 90% CI 1-sided [lower limit -1.2], Standard Deviation 3.9

13. Secondary Outcome: App Usage Behavior
Description: Usage behavior is defined as the proportion of days the app was opened across the 4-month trial period
Time Frame: from baseline through Month 4 (daily)
Population: ITT population: all randomized participants who started the intervention and who had at least one app usage data point. Participants included underactive older adults who own a smartphone.
Measure: Mean (Standard Deviation); unit: proportion of days
Arm/Group | Proof Positive On | Proof Positive Off | Coach Me On | Coach Me Off | On Your Feet On | On Your Feet Off
Number analyzed (Participants) | 54 | 51 | 51 | 54 | 52 | 53
proportion of days | 0.73 (0.28) | 0.68 (0.29) | 0.71 (0.29) | 0.71 (0.28) | 0.68 (0.30) | 0.73 (0.27)
Statistical Analysis 1: Comparison: Proof Positive On vs Proof Positive Off; Test type: Superiority; p = .84, t-test, 2 sided
Statistical Analysis 2: Comparison: Coach Me On vs Coach Me Off; Test type: Superiority; p = .96, t-test, 2 sided
Statistical Analysis 3: Comparison: On Your Feet On vs On Your Feet Off; Test type: Superiority; p = .41, t-test, 2 sided

14. Secondary Outcome: Perceived App Quality (uMARS)
Description: The Mobile App Rating Scale User Version (uMARS) was used to measure user satisfaction with the app, particularly participant's ratings for app quality. The uMARS includes a usability feedback subindex which is comprised of the average of item responses for 4 subsections (engagement, functionality, aesthetics, information), to yield a total quality score. Ratings are on a scale of 1 (low perceived quality, min) to 5 (high perceived quality, max).
Time Frame: 4 months
Population: ITT population: all randomized participants who had valid questionnaire data at post-test. Participants included underactive older adults who own a smartphone.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Proof Positive On | Proof Positive Off | Coach Me On | Coach Me Off | On Your Feet On | On Your Feet Off
Number analyzed (Participants) | 49 | 47 | 46 | 50 | 48 | 48
score on a scale | 3.8 (0.5) | 4.0 (0.6) | 3.9 (0.5) | 4.0 (0.5) | 4.0 (0.5) | 3.9 (0.5)
Statistical Analysis 1: Comparison: Proof Positive On vs Proof Positive Off; Test type: Superiority; p = .13, t-test, 2 sided
Statistical Analysis 2: Comparison: Coach Me On vs Coach Me Off; Test type: Superiority; p = 0.20, t-test, 2 sided
Statistical Analysis 3: Comparison: On Your Feet On vs On Your Feet Off; Test type: Superiority; p = 0.39, t-test, 2 sided

15. Other Pre Specified Outcome: Correlation of Change in Daily Steps to Change in Hypothesized Mediators
Description: Spearman Correlation coefficients were calculated to assess correlations between change in the primary outcome (change in daily steps) and change in hypothesized mediators (i.e., Self-efficacy for Physical Activity Change, Self-regulation of Physical Activity Change, Family Social Support for Physical Activity Change, Outcome Expectation for Physical Activity Change, Aging Self-perceptions (Attitude Toward Own Aging) Change, Views of Aging--Psychosocial Loss Change, Views of Aging--Physical Change Change, Views of Aging--Psychological Growth Change).
Time Frame: baseline to Month 4 change
Population: ITT population: all randomized subjects who started the intervention and had both pre- and post-test values were considered for analyses. Missing values were excluded pairwise within the correlation matrix (i.e., If a data point was missing from either a hypothesized mediator (e.g., family social support for physical activity) OR from activity monitor steps data, then the subject's data point was not included in that particular correlational analysis. Data points available range n=91 to n=96.
Measure: Median (Full Range); unit: change in daily steps
Groups:
- Total Participants: All participants who participated in the study and who had baseline and follow-up measures for each of the given variables. The group includes participants who received various combinations of the Moving Up app specialty feature interventions (Coach Me, On Your Feet, Proof Positive). The total ITT group consists of 105 participants but number of observable data depend on the individual variables within the correlation matrix.
Arm/Group | Total Participants
Number analyzed (Participants) | 96
change in daily steps
  Self-efficacy for Physical Activity Change | -4.8 [-57.8 to 50.0]
  Self-regulation of Physical Activity Change | 0.8 [-0.8 to 4.0]
  Family Social Support for Physical Activity Change: number analyzed (Participants) | 92
  Family Social Support for Physical Activity Change | 0.1 [-3.3 to 3.9]
  Outcome Expectation for Physical Activity Change: number analyzed (Participants) | 92
  Outcome Expectation for Physical Activity Change | 0.0 [-12.8 to 15.4]
  Aging Self-perceptions (Attitude Toward Own Aging) Change | 0.0 [-3.0 to 3.0]
  Views of Aging--Psychosocial Loss Change: number analyzed (Participants) | 95
  Views of Aging--Psychosocial Loss Change | 0.0 [-22.0 to 10.0]
  Views of Aging--Physical Change Change: number analyzed (Participants) | 91
  Views of Aging--Physical Change Change | 0.0 [-15.0 to 13.0]
  Views of Aging--Psychological Growth Change: number analyzed (Participants) | 94
  Views of Aging--Psychological Growth Change | 0.0 [-10.0 to 8.0]
Statistical Analysis 1: Comparison: Total Participants; Correlation between Self-efficacy for Physical Activity change and Daily Steps change across 4 months; Test type: Other; p = 0.3116, t distribution with n-2 degrees of freed; Spearman Correlation = -0.10435
Statistical Analysis 2: Comparison: Total Participants; Correlation between Correlation between Self-regulation of Physical Activity change and Daily Steps change across 4 months; Test type: Other; p = 0.0838, t distribution with n-2 degrees of freed; Spearman Correlation = 0.17742
Statistical Analysis 3: Comparison: Total Participants; Correlation between Family Social Support for Physical Activity change and Daily Steps change across 4 months; Test type: Other; p = 0.3510, t distribution with n-2 degrees of freed; Spearman Correlation = -0.09834
Statistical Analysis 4: Comparison: Total Participants; Correlation between Outcome Expectation for Physical Activity change and Daily Steps change across 4 months; Test type: Other; p = 0.6659, t distribution with n-2 degrees of freed; Spearman Correlation = -0.04562
Statistical Analysis 5: Comparison: Total Participants; Correlation between Aging Self-perceptions (Attitude Toward Own Aging) change and Daily Steps change across 4 months; Test type: Other; p = 0.6402, t distribution with n-2 degrees of freed; Spearman Correlation = -0.04831
Statistical Analysis 6: Comparison: Total Participants; Correlation between Views of Aging--Psychosocial Loss change and Daily Steps change across 4 months; Test type: Other; p = 0.2048, t distribution with n-2 degrees of freed; Spearman Correlation = 0.13128
Statistical Analysis 7: Comparison: Total Participants; Correlation between Views of Aging--Physical Change change and Daily Steps change across 4 months; Test type: Other; p = 0.3445, t distribution with n-2 degrees of freed; Spearman Correlation = 0.10022
Statistical Analysis 8: Comparison: Total Participants; Correlation between Views of Aging--Psychological Growth change and Daily Steps change across 4 months; Test type: Other; p = 0.9340, t distribution with n-2 degrees of freed; Spearman Correlation = -0.00866

ADVERSE EVENTS:
Time Frame: Adverse events were reported to the PI within 24 hours of their occurrence across the 4-month trial.
Description: All potential adverse events were reported to the PI to determine reporting to the USC IRB.
Arm/Group | AT App + On Your Feet+ CoachMe+ Proof Pos | AT App + On Your Feet + Coach Me | AT App + On Your Feet + Proof Positive | AT App + On Your Feet | AT App + Coach Me + Proof Positive | AT App + Coach Me | AT App + Proof Positive | AT App
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/13 | 0/13 | 0/14 | 0/14 | 0/12 | 0/15 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13 | 0/13 | 0/14 | 0/14 | 0/12 | 0/15 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/13 | 0/13 | 0/14 | 0/14 | 1/12 | 0/15 | 0/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AT App + On Your Feet+ CoachMe+ Proof Pos (N=12) | AT App + On Your Feet + Coach Me (N=13) | AT App + On Your Feet + Proof Positive (N=13) | AT App + On Your Feet (N=14) | AT App + Coach Me + Proof Positive (N=14) | AT App + Coach Me (N=12) | AT App + Proof Positive (N=15) | AT App (N=12)
Excessive weight loss (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Weight loss is beyond that which is expected for changes in physical activity over a four-month period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-09): https://cdn.clinicaltrials.gov/large-docs/40/NCT03417440/Prot_SAP_001.pdf
  • Informed Consent Form (2020-03-23): https://cdn.clinicaltrials.gov/large-docs/40/NCT03417440/ICF_000.pdf